CLINICAL TRIAL: NCT05580900
Title: California Fatherhood: Family-Focused, Interconnected, Resilient, and Essential (Cal-FIRE)
Brief Title: Evaluating How Course Modality Influences the Effectiveness of the R3 Academy for Dads
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthy Relationships California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 90ZJ0046
Record Dates: First submitted 2022-09-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Program Modality
Keywords: Fatherhood Program; modality; evaluation; father; comparison; propensity score matching; live; in-person; livestream; online
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: In our quasi-experimental design, we allow participants to select whether they want to participate in a live or livestream program modality. The fatherhood curriculum is the same for both, only the mode of delivery is different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Livestream Modality (Experimental): The livestream modality is considered the treatment group for the purpose of this quasi-experimental study.
  Interventions: Other: Livestream Modality (treatment)
- Live Modality (Experimental): The live modality is considered the control group for the purpose of this quasi-experimental study.
  Interventions: Other: Live Modality (control)

INTERVENTIONS:
Other: Livestream Modality (treatment) — For this evaluation, the livestream modality is considered the treatment.
  Arms: Livestream Modality
Other: Live Modality (control) — For this evaluation, the live or in-person modality is considered the control group.
  Arms: Live Modality

SUMMARY:
The Cal-FIRE project is designed to offer the R3 Academy for Dads, a robust 24-hour program, to predominantly low-income adult fathers, ages 18 and over in the state of California. The R3 Academy is an evidence-based parenting curriculum that helps fathers strengthen their relationships with their child, with their spouse/co-parent, and at work. The program also includes two evidence-based components that address economic stability and an innovative approach to Case Management that fosters client self-direction. The R3 Academy curricula will be delivered in both English and Spanish through two modalities: 1) live classes and 2) livestream classes via a video conferencing platform. The Local Evaluation will examine how modality, or in other words attending a live class versus a livestream class, influences the effectiveness of responsible fatherhood education when it comes to father involvement and coparenting. The question of modality is a timely one. In the COVID-19 era, many programs have become exclusively online-but the potential impact on effectiveness is not well known. Data from this study will help illuminate what can be gained or jeopardized in a world increasingly moving toward modes of virtual engagement. Specifically, the current evaluation will explore potential similarities and differences related to the implementation of the two modalities and their influence of father outcomes. Specific research questions include:

RQ1: How do live (control) and livestream (treatment) responsible fatherhood workshops compare on father involvement outcomes? RQ2: How do live (control) and livestream (treatment) workshops compare on father involvement outcomes? RQ3: Do program effects last beyond program completion?

DETAILED DESCRIPTION:
Fathers in this study are required to take an Eligibility survey. If they meet the required eligibility criteria, the survey will gather further information including screening factors associated with domestic violence that, if checked, will be flagged for further assessment by personal contact with our Case Management Supervisor. This form also will enable the registrant to identify which class format he wishes to attend-a live R3 Academy or a livestream workshop via a video conferencing platform. For the purpose of this study, the live or in-person modality is considered the control group and the livestream workshop is considered the treatment group. The R3 Academy curriculum is the same for each group, only the modality of curriculum delivery is different. Courses are a total of 24 hours and are split into either 6- or 12-week formats. Incentives for program completion include a $50 gift card that is offered to those who complete at least 90% of the program. In addition to the Eligibility survey, participants are asked to take a pre-survey before starting the class, a post-survey immediately following class completion, and a 4-month follow-up survey. If participants complete all three surveys they are eligible for an additional $25 gift card which they can receive even if they did not reach 90% completion.

As stated previously, entry into treatment or control groups is determined at enrollment. At the time of the impact analysis, propensity score matching (PSM) comparison groups will be formed-this statistical analysis will match up similar participants from each group to allow for comparison across conditions. PSM allows researchers to estimate differences between treatment and control groups in non-randomized samples. PSM will allow us to directly compare matched cases-meaning that the treatment and control groups will have a similar distribution of sociodemographic and sociocultural characteristics. This allows us to consider how outcomes vary between treatment and control groups, while accounting for the potential self-selection into different program groups. Participants will be matched across multiple metrics, including: racial/ethnic identity, sex/gender, income, education level, language of instruction, number of children, employment status, age, marital status, and residential status. As clients may choose one program delivery modality over another due to work, childcare availability, or time, measures will be included for work schedule, availability of social support, work flexibility, and work-family stress.

ELIGIBILITY:
Inclusion Criteria:

* Fathers have to be at least 18 years old with at least one child 24 years old or younger and residing in California.

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Fathers
Enrollment: 510 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Father Involvement after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion which can be 6 to 12 weeks after baseline depending on the class attended, and (3) 4 months after course completion.
  The Fatherhood Research & Practice Network Father Engagement Scale is broken down into two subscales: father caregiving and father support. The father caregiving inquired how frequently fathers participate in a list of activities such as feeding, caring for, or playing with their child. The father support subscale asked how often father participated in activities such as encouraging and talking to their children. Responses are given on a 0=Never to 4=Every day Likert scale.
Changes in father's Coparenting after program completion and 4 months following program completion | Data is collected at three time points: (1) before attending the class, (2) immediately after class completion which can be 6 to 12 weeks after baseline depending on the class attended, and (3) 4 months after course completion.
  The Fatherhood Research & Practice Network Coparenting Scale is a 10 item scale where father were asked a series of questions related to their coparenting relationships. Answers ranged from 0=strongly disagree to 4=strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shafer, PhD, Principal Investigator — Brigham Young University; Jason Krafsky, Study Director — Healthy Relationships California; Patty Howell, Study Chair — Healthy Relationships California; Dyann Collins, Study Chair — Healthy Relationships California
Locations (1):
- Healthy Relationships California, Leucadia, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be archived with the Inter-university Consortium for Political and Social Research (ICPSR) after we complete our research. The data will not include the participant's name, address, date of birth, phone number, or any other personal information or ID numbers that could identify the participant. Archiving this data provides other researchers with the opportunity to learn about how relationship education benefits people. Information about data archival will be provided on the consent form.